CLINICAL TRIAL: NCT04383873
Title: Effectiveness Analysis of Armeo Spring Device as a Rehabilitation Treatment in Spinal Cord Injured Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Nacional de Parapléjicos de Toledo (Other)
Responsible Party: Principal Investigator, Ana de los Reyes Guzmán, Principal Investigator, Hospital Nacional de Parapléjicos de Toledo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C501/2016
Record Dates: First submitted 2020-04-20; First posted 2020-05-12 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Spinal Cord Injury Cervical
Keywords: Effectiveness; Rehabilitation; Upper extremity; Spinal Cord Injury cervical; Robotic device

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 17 cervical Spinal Cord injured patients daily receive 1 hour of upper extremity therapy
  Interventions: Device: Training by means of Armeo Spring device; Other: Current treatment based on conventional therapy
- Control (Active Comparator): 17 cervical Spinal Cord injured patients daily receive 1 hour of upper extremity therapy
  Interventions: Other: Current treatment based on conventional therapy; Other: Additional treatment based on conventional therapy

INTERVENTIONS:
Device: Training by means of Armeo Spring device — This patients group receive 40 experimental sessions. Each session is based on 30 min by using Armeo Spring device.
  Arms: Intervention
Other: Current treatment based on conventional therapy — All the patients enrollment in the study receive 30 min of conventional therapy during 40 sessions.
Other: Additional treatment based on conventional therapy — This intevention was added for providing the same amount of therapy than those patients randomly enrolled in the intervention group. So, patients in the control group receive other 30 min of conventional therapy added on current treatment during 40 sessions.
  Arms: Control

SUMMARY:
Loss of motor function is a consequence after a spinal cord injury (SCI). The incidence of SCI varies greatly from 12.1 to 57.8 cases per million depending on the country. More than 50% of people with SCI have impaired upper limb (UL) function, experiencing limitations in performing functional tasks. In this context, one of the rehabilitation objectives is to achieve the maximum level of independence in the patient in the performance of activities of daily living (ADL).

Within the clinical setting, the main motivation in the use of robotic devices and/or exoskeletons for a rehabilitation purpose focuses on the fact that these help therapists in administering repetitive manual therapies to patients during exercises. There is evidence that the amount of therapy patients receive is insufficient. Without creating additional time demands on clinicians, robotic devices can perform the repetitive mechanical aspects of therapy, increasing the amount of therapy that patients receive. However, the current evidence in stroke patients suggests that the improvements observed are due to the intensity of the therapy, regardless of whether the administration of rehabilitation is due to robotic devices and/or traditional means.

The main objective of this study is to analyze the effectiveness of the commercial Armeo® Spring system (Hocoma AG, Switzerland) and a Virtual Reality application to repeatedly work the ADL from drinking from a glass, in people with cervical SCI. The ADL of drinking has been chosen, as a representative activity of those related to food, which requires control, strength and coordination of the UL. The study is carried out at the Hospital Nacional de Parapléjicos with the collaboration of Occupational Therapy Unit, the Rehabilitation Department, and the Biomechanics and Technical Aids Unit. This effectiveness is measured in terms of functional improvements and in the quality of the UL movements performed.

DETAILED DESCRIPTION:
In the literature, there are several studies of the upper limb applied to ADL. The analysis of complete ADL is related to the clinical objectives of the rehabilitative treatment of the UL. An important part of rehabilitation after neurological injuries consists of training activities aimed at fulfilling a function or objective, in which patients have to move their arms continuously repeating certain movement patterns. This is currently one of the main strategies to promote recovery of upper limb function in people who have suffered a spinal cord injury (SCI) o stroke.

Within the clinical setting, the main motivation in the use of robotic devices and/or exoskeletons for a rehabilitation purpose focuses on the fact that these help therapists in administering repetitive manual therapies to patients during exercises. There is evidence that the amount of therapy patients receive is insufficient. Without creating additional time demands on clinicians, robotic devices can perform the repetitive mechanical aspects of therapy, increasing the amount of therapy that patients receive. On the other hand, the use of robotic devices is closely linked to the use of virtual reality (VR) applications. VR interfaces provide feedback to the patient, increasing their level of motivation and adherence to the task during therapy. In this way, therapies with robotic devices and / or exoskeletons increase the amount of rehabilitation, the level of motivation of the patient, and training oriented to fulfill a function or task. Rehabilitation of patients with robotic device-based therapies in addition to traditional therapies could improve functional outcomes. However, the current evidence in stroke patients suggests that the improvements observed are due to the intensity of the therapy, regardless of whether the administration of rehabilitation is due to robotic devices and/or traditional means.

The main objective of this study is to analyze the effectiveness of the commercial Armeo® Spring system (Hocoma AG, Switzerland) and a Virtual Reality application to repeatedly work the ADL from drinking from a glass, in people with cervical SCI. The ADL of drinking has been chosen, as a representative activity of those related to food, which requires control, strength and coordination of the UL. The study is carried out at the Hospital Nacional de Parapléjicos with the collaboration of Occupational Therapy Unit, the Rehabilitation Department, and the Biomechanics and Technical Aids Unit. This effectiveness is measured in terms of functional improvements and in the quality of the UL movements performed.

The secondary objectives are:

* To validate the applicability of the Virtual Reality developed to work the upper limb during the execution of a complete AVD.
* To know the usability and level of acceptance of this therapy in patients with spinal cord injury and UL functional impairments.
* To quantify the differences between the functional patterns of both groups, intervention and control, by means of objective measures, functional scales and measures of the quality of movement, collected in patient evaluations, before, during and after treatment.
* To determine the influence of the RV and the Armeo Spring exoskeleton on the motor recovery of patients with spinal cord injury and UL impairments.

ELIGIBILITY:
Inclusion Criteria:

* Cervical lesions above C8, incomplete in the motor aspect or complete with zones of partial motor preservation at least C6, classified according to the ASIA scale.
* Traumatic or non-progressive medical etiology.
* Less than 6 months of injury evolution (subacute).
* Age between 16 and 75 years.
* To have reached the seated posture.
* Be informed and consent to participate in the study.

Exclusion Criteria:

* Unstable orthopaedic injuries such as unconsolidated fractures or with unstable osteosynthesis systems in upper limbs.
* Skin lesions and/or pressure ulcers in the exoskeleton placement area.
* Having joint stiffness and/or severe spasticity.
* Bronchopneumopathy and/or severe heart disease that will require monitoring during exercise.
* Visual problems.
* Cognitive impairment.
* Do not sign the corresponding informed consent.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-06-18 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Clinical scale SCIM | At baseline
  The Spinal Cord Independence Measure (SCIM) is a new disability scale developed specifically for patients with spinal cord lesions in order to make the functional assessments of patients with paraplegia or tetraplegia more sensitive to changes. Exclusively designed for spinal injury. It consists of 3 subscales. The total score varies from 0-100 points, where 0 corresponds to the highest degree of dependency and 100 to the highest degree of independence.
Change from baseline Clinical scale SCIM at 10 weeks | At the end of the study (at week 10)
  The Spinal Cord Independence Measure (SCIM) is a new disability scale developed specifically for patients with spinal cord lesions in order to make the functional assessments of patients with paraplegia or tetraplegia more sensitive to changes. Exclusively designed for spinal injury. It consists of 3 subscales. The total score varies from 0-100 points, where 0 corresponds to the highest degree of dependency and 100 to the highest degree of independence.
Clinical scale CUE | At baseline
  Capabilities of Upper Extremity (CUE) measures upper extremity functional limitations in individuals with tetraplegia. The patient reports the outcome about how well you are able to use the arms and hands of patients. 32 item questionnaire with items in 7 domains. Self-reported measure performed by interview.
  Score on 7 points scale representing self-perceived difficulty: 1 (Totally limited, can´t do at all) y 7 (Not at all limited). So, the minimum score is 32 (worse result) and the maximum score 224 (greater function)
Change from baseline Clinical scale CUE at 10 weeks | At the end of the study (at week 10)
  Capabilities of Upper Extremity (CUE) measures upper extremity functional limitations in individuals with tetraplegia. The patient reports the outcome about how well you are able to use the arms and hands of patients. 32 item questionnaire with items in 7 domains. Self-reported measure performed by interview.
  Score on 7 points scale representing self-perceived difficulty: 1 (Totally limited, can´t do at all) y 7 (Not at all limited). So, the minimum score is 32 (worse result) and the maximum score 224 (greater function)
Clinical Scale Jebsen-Taylor Hand Function (JTHF) | At baseline
  The Jebsen-Taylor function test was designed to provide a short, objective test of hand functions commonly used in activities of daily living (ADLs). The target patient population includes adults with neurological or musculoskeletal conditions involving hand disabilities, although there may be other patient populations with other hand dysfunctions which may be appropriate. It consists of seven items that include a range of fine motor, weighted and non-weighted hand function activities which are timed: writing (copying) a 24-letter sentence turning over a 3 × 5" cards, picking up small common objects such as a coin and bottle cap, simulated feeding using a teaspoon and five kidney beans, stacking checkers picking up large light objects such as an empty tin can, and picking up and moving large weighted cans. The scale measures the time in seconds in reaching each task. A higher spent time is a worse outcome.
Change from baseline Clinical Scale Jebsen-Taylor Hand Function (JTHF) at 10 weeks | At the end of the study (at week 10)
  The Jebsen-Taylor function test was designed to provide a short, objective test of hand functions commonly used in activities of daily living (ADLs). The target patient population includes adults with neurological or musculoskeletal conditions involving hand disabilities, although there may be other patient populations with other hand dysfunctions which may be appropriate. It consists of seven items that include a range of fine motor, weighted and non-weighted hand function activities which are timed: writing (copying) a 24-letter sentence turning over a 3 × 5" cards, picking up small common objects such as a coin and bottle cap, simulated feeding using a teaspoon and five kidney beans, stacking checkers picking up large light objects such as an empty tin can, and picking up and moving large weighted cans. The scale measures the time in seconds in reaching each task. A higher spent time is a worse outcome.
Clinical scale Nine Hole Peg Test | At baseline
  The Nine-Hole Peg Test (9-HPT) is a standardized, quantitative assessment used to measure finger dexterity. The scale measures the time in seconds in reaching each task. A higher spent time is a worse outcome.
Change from baseline Clinical scale Nine Hole Peg Test at 10 weeks | At the end of the study (at week 10)
  The Nine-Hole Peg Test (9-HPT) is a standardized, quantitative assessment used to measure finger dexterity. The scale measures the time in seconds in reaching each task. A higher spent time is a worse outcome.
Clinical Scale GRASSP | At baseline
  The GRASSP is a clinical impairment measure specific to the upper limb for use after tetraplegia. The GRASSP measure sensorimotor and prehension function through three domains, important in describing arm and hand function: Strength, Sensation, Prehension. The minimal score is 0 (worse outcome) and the maximum 98 (better outcome) for each hand.
Change from baseline Clinical Scale GRASSP at 10 weeks | At the end of the study (at week 10)
  The GRASSP is a clinical impairment measure specific to the upper limb for use after tetraplegia. The GRASSP measure sensorimotor and prehension function through three domains, important in describing arm and hand function: Strength, Sensation, Prehension. The minimal score is 0 (worse outcome) and the maximum 98 (better outcome) for each hand.
Edinburg Handedness Test | At baseline
  Most people are right handed. The Edinburgh Handedness Inventory is a well known short questionnaire for determining objectively whether one is left or right handed and there is a short form of it. 10 items are valued. The total score is 50 points and the minimum 10 points. The closer score to 50 points, more left-handed the person is. And the closer score to 10 the more right-handed.
Kinematic indices | At baseline
  This assessment is performed by means of photogrammetry. Markers are placed on the trunk and the arm analyzed, and kinematic variables about the UL movement are computed in terms of accuracy, agility, coordination, efficiency and smoothness. A score of 100 in each index corresponds to the healthy pattern. The minimun and worse outcome is 0 score.
Change from baseline Kinematic indices at 10 weeks | At the end of the study (at week 10)
  This assessment is performed by means of photogrammetry. Markers are placed on the trunk and the arm analyzed, and kinematic variables about the UL movement are computed in terms of accuracy, agility, coordination, efficiency and smoothness. A score of 100 in each index corresponds to the healthy pattern. The minimun and worse outcome is 0 score.

SECONDARY OUTCOMES:
Compliance | At the end of the study (at week 10)
  The total sessions number that the patient has performed and the duration in weeks
QUEST usability scale | At the end of the study (at week 10)
  At ending the treatment using Armeo Spring, patients show their opinion and satisfaction level with the experimental scenario
TMS assessment | At baseline
  A transcranial magnetic stimulation-based assessment is made.
Change from baseline TMS assessment at 10 weeks | At the end of the study (at week 10)
  A transcranial magnetic stimulation-based assessment is made.
Beck's Depression Inventory | At baseline
  This depression inventory can be self-scored. The scoring scale is at the end of questionnaire. the BDI consists of 21 items, self-reporting inventory for assessing depression, with 4 alternatives each that are rated from 0 to 3, giving a possible total of 0 to 63 points. The interpretation of the score is as follows: From 1-10 points: These ups and downs are considered normal; from 11-16 points: Slight disturbance of mood; from 17-20 points: Intermittent states of depression. From 21-30 points: Moderate depression. 31-40 points: Severe depression; More than 40 points: Extreme depression.
Change from baseline Beck's Depression Inventory at 10 weeks | At the end of the study (at week 10)
  This depression inventory can be self-scored. The scoring scale is at the end of questionnaire. the BDI consists of 21 items, self-reporting inventory for assessing depression, with 4 alternatives each that are rated from 0 to 3, giving a possible total of 0 to 63 points. The interpretation of the score is as follows: From 1-10 points: These ups and downs are considered normal; from 11-16 points: Slight disturbance of mood; from 17-20 points: Intermittent states of depression. From 21-30 points: Moderate depression. 31-40 points: Severe depression; More than 40 points: Extreme depression.
Hospital Anxiety and Depression Scale (HADS) | At baseline
  The HADS is a questionnaire widely used to evaluate the anxiety and depression. The HADS takes between 2 to 5 minutes to complete. The HAD contains seven subscales for each mood (anxiety and depression). The HAD Scale is an effective screening instrument and ranges of scores are given in order that the proportion of false positives or false negatives may be minimized. Regarding the scores obtained, a score equal to or greater than 11 is considered depression/anxiety. Between 0 and 7 is not considered depression/anxiety, and between 8 and 10 is doubtful case.
Change from baseline Hospital Anxiety and Depression Scale (HADS) at 10 weeks | At the end of the study (at week 10)
  The HADS is a questionnaire widely used to evaluate the anxiety and depression. The HADS takes between 2 to 5 minutes to complete. The HAD contains seven subscales for each mood (anxiety and depression). The HAD Scale is an effective screening instrument and ranges of scores are given in order that the proportion of false positives or false negatives may be minimized. Regarding the scores obtained, a score equal to or greater than 11 is considered depression/anxiety. Between 0 and 7 is not considered depression/anxiety, and between 8 and 10 is doubtful case.

CONTACTS AND LOCATIONS:
Overall Officials: Ana de los Reyes, PhD, Principal Investigator — Hospital Nacional de Parapléjicos
Locations (1):
- Hospital Nacional de Parapléjicos, Toledo, Spain